CLINICAL TRIAL: NCT00003452
Title: Phase II Study of Antineoplastons A10 and AS2-1 In Patients With Carcinoma of the Bladder
Brief Title: Antineoplastons A10 and AS2-1 In Patients With Carcinoma of the Bladder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066483; BC-BL-02 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Stage IV Bladder Cancer
Keywords: recurrent bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplastons (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Stage IV Bladder Cancer will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for Stage IV bladder cancer provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Stage IV bladder cancer

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Stage IV bladder cancer.

DETAILED DESCRIPTION:
Stage IV bladder cancer patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Stage IV bladder cancer, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Stage IV bladder cancer.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV bladder carcinoma that is unlikely to respond to existing therapy and for which no curative therapy exists or stage IV newly diagnosed, incurable bladder carcinoma
* Measurable disease by CT scan
* Tumor must be greater than 2 cm at the largest diameter for the lymph nodes located in the head, neck, axillary, inguinal, or femoral areas and at least 0.5 cm in the largest diameter for other localizations
* 18 and over
* Karnofsky 60-100%
* Life expectancy: greater than 2 months
* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3
* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure
* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium
* No severe heart disease
* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium
* No severe lung disease
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections or fever
* No other serious concurrent disease
* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* Concurrent corticosteroids allowed
* At least 8 weeks since prior radiotherapy and recovered
* Recovered from any prior operative procedure
* Prior cytodifferentiating agent allowed

Exclusion Criteria:

- Prior antineoplaston therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 1996-05-06 (Actual); Primary Completion 1998-05-04 (Actual); Study Completion 1998-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com